CLINICAL TRIAL: NCT01714635
Title: Clinical Investigation of Expanded Designs of the Tecnis® Multifocal 1-Piece IOL
Brief Title: Clinical Investigation of Expanded Designs of a Multifocal IOL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DIOL-106-ZMLA
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Results first posted 2015-01-15 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2014-11

CONDITIONS: Cataract
Keywords: cataract; IOL; intraocular lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tecnis Multifocal Intraocular lens #1 (Experimental): A low diopter add multifocal intraocular lens
  Interventions: Device: Tecnis Multifocal Intraocular Lens
- Tecnis Multifocal Intraocular Lens #2 (Experimental): A low diopter add multifocal intraocular lens
  Interventions: Device: Tecnis Multifocal Intraocular Lens
- Monofocal Intraocular Lens (Active Comparator): Commercially available monofocal intraocular lens (IOL)
  Interventions: Device: Monofocal Intraocular Lens

INTERVENTIONS:
Device: Tecnis Multifocal Intraocular Lens
  Arms: Tecnis Multifocal Intraocular Lens #2; Tecnis Multifocal Intraocular lens #1
Device: Monofocal Intraocular Lens
  Arms: Monofocal Intraocular Lens

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and effectiveness of the TECNIS Multifocal 1-Piece Intraocular Lens (IOLs), Models ZKB00 and ZLB00 which will each provide statistically better distance-corrected near visual acuity compared to the monofocal control lens. Complication and adverse event rates associated with each Multifocal IOL will be within the ISO SPE rate for posterior chamber IOLs.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years of age
* Bilateral cataracts for which phacoemulsification extraction and posterior IOL implantation have been planned for both eyes
* Preoperative best-corrected distance visual acuity (BCDVA) of 20/40 or worse (Snellen) with or without a glare source
* Potential for postoperative best-corrected visual acuity of 20/25 or better
* Preoperative corneal astigmatism of 1.0 D or less with normal corneal topography and no irregular corneal astigmatism
* Clear intraocular media, other than cataract
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures
* Signed informed consent and HIPAA authorization or equivalent documentation necessary to comply with applicable privacy laws pertaining to medical treatment in the governing countries
* Ability to understand and respond to a questionnaire verbally administered in English

Exclusion Criteria:

* Requiring an intraocular lens power outside the available range of +16.0 to +28.0 D
* Pupil abnormalities (non-reactive, fixed pupils, or abnormally shaped pupils)
* Recent ocular trauma or ocular surgery that is not resolved/stable or may affect visual outcomes
* Prior refractive (LASIK, LASEK, RK, PRK, etc.) or intraocular surgery
* Corneal abnormalities such as stromal, epithelial or endothelial dystrophies that are predicted to cause visual acuity losses to a level of 20/30 or worse during the study
* Inability to achieve keratometric stability for contact lens wearers
* Subjects with diagnosed degenerative visual disorders (e.g., macular degeneration or other retinal disorders) that are predicted to cause visual acuity losses to a level of 20/30 or worse during the study
* Subjects with conditions associated with increased risk of zonular rupture, including capsular or zonular abnormalities that may lead to IOL decentration, including pseudoexfoliation, trauma, or posterior capsule defects
* Use of systemic or ocular medications that may affect vision
* Prior, current, or anticipated use during the course of the 12-month study of tamsulosin or silodosin (e.g., Flomax®, Flomaxtra®, Rapaflo®) likely, in the opinion of the investigator, to cause poor dilation or lack of adequate iris structure to perform standard cataract surgery
* Inability to focus, fixate or maintain binocular vision for prolonged periods of time (e.g., due to strabismus, nystagmus, etc.)
* Poorly-controlled diabetes
* Acute, chronic, or uncontrolled systemic or ocular disease or illness that, in the opinion of the investigator, would increase the operative risk or confound the outcomes of the study (e.g., immunocompromised, connective tissue disease, suspected glaucoma, glaucomatous changes in the fundus or visual field, ocular inflammation, etc.). Note: ocular hypertension without glaucomatous changes is acceptable.
* Known ocular disease or pathology that may affect visual acuity or that may be expected to require retinal laser treatment or other surgical intervention during the course of the study (macular degeneration, cystoid macular edema, diabetic retinopathy, etc.)
* Patient is pregnant, plans to become pregnant, is lactating or has another condition associated with the fluctuation of hormones that could lead to refractive changes
* Concurrent participation or participation within 30 days prior to preoperative visit in any other clinical trial
* Desire for monovision correction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2012-11; Primary Completion 2013-10 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kendra Hileman, PhD, Study Director — Abbott Medical Optics
Locations (18):
- United States (17):
  - Fishkind, Bakewell & Maltzman Eye Care & Surgery Center, Tucson, Arizona
  - Boozman-Hof Regional Eye Clinic, Rogers, Arkansas
  - Empire Eye & Laser Center, Bakersfield, California
  - Assil Eye Institute, Beverly Hills, California
  - Cape Coral Eye Center (Argus Research Center), Cape Coral, Florida
  - Virdi Eye Clinic & Laser Vision Center, Rock Island, Illinois
  - Eye Surgeons of Indiana, Indianapolis, Indiana
  - Wallace Eye Surgery, Alexandria, Louisiana
  - Pepose Vision Institute, Chesterfield, Missouri
  - Ophthalmic Consultants of Long Island, Rockville Centre, New York
  - The Eye Center of Central PA, Allenwood, Pennsylvania
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Bucci Cataract & Laser Vision, Wilkes-Barre, Pennsylvania
  - Loden Vision Center, Goodlettsville, Tennessee
  - Whitsett Vision Group, Houston, Texas
  - Lone Star Eye Care, Sugar Land, Texas
  - Clarus Eye Centre, Lacey, Washington
- The Midline Eye Institute, Solihull, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Tecnis Multifocal Intraocular Lens #1; Tecnis Multifocal Intraocular Lens #2: A low diopter add multifocal intraocular lens
  Tecnis Multifocal Intraocular Lens
- Monofocal Intraocular Lens: Commercially available monofocal intraocular lens (IOL)
  Monofocal Intraocular Lens
Period: Overall Study
Arm/Group | Tecnis Multifocal Intraocular Lens #1 | Tecnis Multifocal Intraocular Lens #2 | Monofocal Intraocular Lens
Started | 147 | 150 | 148
Completed | 145 | 150 | 146
Not Completed | 2 | 0 | 2
Not completed — Discontinued | 1 | 0 | 2
Not completed — Missed 6-month exam | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tecnis Multifocal Intraocular Lens #1 | Tecnis Multifocal Intraocular Lens #2 | Monofocal Intraocular Lens | Total
Number analyzed (Participants) | 147 | 150 | 148 | 445
Age, Customized [Number; unit: participants] — Age was grouped by catagories as described in the table.
  participants
    Less than 60 years | 21 | 18 | 13 | 52
    60 - 69 years | 58 | 68 | 67 | 193
    70 - 79 years | 66 | 59 | 60 | 185
    Greater than or equal to 80 years | 2 | 5 | 8 | 15
    Not reported | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 101 | 85 | 260
  Male | 73 | 49 | 63 | 185
Region of Enrollment [Number; unit: participants]
  United States | 146 | 150 | 147 | 443
  United Kingdom | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Monocular Distance-corrected Near Visual Acuity (VA) at 40 cm
Description: Mean (LogMAR) monocular distance-corrected near VA at 40 cm at six months postoperative
Time Frame: six months
Population: eyes
Measure: Mean (Standard Deviation); unit: LogMAR VA
Arm/Group | Tecnis Multifocal Intraocular Lens #1 | Tecnis Multifocal Intraocular Lens #2 | Monofocal Intraocular Lens
Number analyzed (Participants) | 147 | 150 | 148
LogMAR VA | 0.253 (0.012) | 0.179 (0.011) | 0.582 (0.014)

2. Secondary Outcome: Mean Diopter Range With VA of 20/40 or Better
Description: Mean diopter range in which VA of 20/40 or better was achieved at six months. Note: diopter range outcome measure was obtained from a substudy group that included the first 10 study sites to reach enrollment goals. Among these 10 sites, the first 60 subjects in each lens group (approximately*) to reach the 6-month visit were included in the substudy.
  * The intent was to enroll 60 subjects per group, but group #1, group #2, and the monofocal group had 59, 63, and 61 subjects, respectively.
Time Frame: six months
Population: eyes
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Tecnis Multifocal Intraocular Lens #1 | Tecnis Multifocal Intraocular Lens #2 | Monofocal Intraocular Lens
Number analyzed (Participants) | 59 | 63 | 61
diopters | 3.16 (0.50) | 3.30 (0.69) | 1.75 (0.70)

3. Secondary Outcome: Spectacle Independence
Description: Number of subjects never requiring spectacles at six months. This outcome measure was obtained via questionnaire. The questionnaire was administered by phone.
Time Frame: six months
Population: Five subjects (3 from Group #1 [145-142], 1 from Group #2 [150-149], and 1 from the monofocal control group [146-145]) did not complete the questionnaire because they were unavailable, refused to complete it, implant status precluded completion (bilateral implants required), or failed to answer this particular question.
Measure: Number; unit: participants
Arm/Group | Tecnis Multifocal Intraocular Lens #1 | Tecnis Multifocal Intraocular Lens #2 | Monofocal Intraocular Lens
Number analyzed (Participants) | 142 | 149 | 145
participants | 87 | 111 | 3

ADVERSE EVENTS:
Arm/Group | Tecnis Multifocal Intraocular Lens #1 | Tecnis Multifocal Intraocular Lens #2 | Monofocal Intraocular Lens
Serious Adverse Events (participants affected / at risk) | 2/147 | 8/150 | 3/148
Other Adverse Events (participants affected / at risk) | 0/147 | 0/150 | 0/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tecnis Multifocal Intraocular Lens #1 (N=147) | Tecnis Multifocal Intraocular Lens #2 (N=150) | Monofocal Intraocular Lens (N=148)
Secondary surgical intervention - not lens-related (Eye disorders) | 0 (0) | 4 (5) | 1 (1)
Secondary surgical intervention - lens-related (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Orbital fracture (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — Orbital fracture was attributed to a fall. Subject also sustained limbal wound rupture and iris prolapse.
Central retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Endophthalmitis/hypopyon (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cystoid macular edema (Eye disorders) | 2 (2) | 0 (0) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the trial is completed, investigators must obtain approval from AMO in writing prior to disclosing trial results.